CLINICAL TRIAL: NCT07335666
Title: Virtual Reality Versus Distraction Game Cards for Reducing Fear, Anxiety, Pain, and Physiological Stress During Pediatric Open Wound Care
Brief Title: Virtual Reality Outperforms Game Card Distraction in Reducing Distress During Pediatric Wound Care
Acronym: VR-WOUND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR-WOUNDCARE-04
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Wounds; Procedural Pain; Procedure-Related Anxiety; Procedural Fear
Keywords: Virtual Reality; Distraction Techniques; Game Card Distraction; Immersive Distraction; Pediatric Wound Care; Child-Centered Care; Pediatric Anxiety; Non-Pharmacological Intervention; Procedural Pain Management
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1:1 ratio to one of three parallel groups: standard care alone (control), standard care with distraction game cards, or standard care with immersive virtual reality glasses.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the distraction interventions, participants and care providers were not blinded. Outcome assessment and data entry were performed by a research assistant who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care Control Group (No Intervention): Participants received standard pediatric wound care according to institutional protocols, including wound cleansing, debridement, suturing when clinically indicated, and dressing application, without any structured distraction intervention.
- Distraction Game Card Group (Experimental): Participants received standard wound care combined with distraction using illustrated game cards. Children engaged in visual search and pattern recognition activities facilitated by a trained researcher throughout the wound care procedure.
  Interventions: Behavioral: Distraction Game Cards
- Virtual Reality Distraction Group (Experimental): Participants received standard wound care combined with immersive virtual reality distraction delivered through virtual reality glasses displaying age-appropriate three-dimensional and 360-degree content during the procedure.
  Interventions: Behavioral: Virtual Reality Distraction

INTERVENTIONS:
Behavioral: Distraction Game Cards — Laminated illustrated game cards containing visual search and pattern-recognition tasks were used as a behavioral distraction during pediatric wound care. A trained researcher facilitated engagement by asking structured questions approximately every 15-30 seconds throughout the procedure to maintain the child's attention.
  Arms: Distraction Game Card Group
Behavioral: Virtual Reality Distraction — Immersive virtual reality distraction was delivered using virtual reality glasses connected to a smartphone displaying age-appropriate three-dimensional and 360-degree audiovisual content throughout the wound care procedure to provide multisensory engagement and reduce procedural distress.
  Arms: Virtual Reality Distraction Group

SUMMARY:
Children often experience fear, anxiety, and pain during wound care procedures, which can make treatment more difficult and distressing. Non-pharmacological distraction techniques may help reduce these negative experiences without the use of medications. Virtual reality (VR) provides immersive visual and auditory stimulation, while simple distraction tools such as game cards offer a low-cost alternative.

This randomized controlled study aims to compare the effectiveness of immersive virtual reality glasses and distraction game cards in reducing fear, anxiety, pain, and physiological stress responses in children aged 5 to 10 years undergoing open wound care. Ninety children are randomly assigned to one of three groups: standard care alone, standard care with distraction game cards, or standard care with virtual reality glasses. Psychological outcomes (fear, anxiety, and pain) and physiological indicators (heart rate and oxygen saturation) are measured before and after the wound care procedure. The results of this study will help identify effective, non-pharmacological strategies to improve children's experiences during painful medical procedures and support child-centered care in pediatric clinical settings.

DETAILED DESCRIPTION:
Open wound care procedures are common in pediatric emergency settings and are frequently associated with fear, anxiety, pain, and physiological stress in children. These responses may interfere with cooperation during treatment and negatively affect children's short- and long-term perceptions of healthcare. Although pharmacological approaches can reduce pain, non-pharmacological interventions are increasingly recommended as complementary strategies to minimize distress without additional medical risk.

Distraction techniques represent one of the most widely used non-pharmacological approaches in pediatric care. Immersive virtual reality (VR) has gained attention as a promising distraction method due to its ability to provide multisensory engagement and strong attentional capture. By immersing children in an interactive virtual environment, VR may reduce awareness of painful stimuli and procedural threat. In contrast, distraction game cards offer a simple, low-cost alternative that engages children cognitively through visual search and pattern recognition tasks. Despite growing evidence supporting both approaches, direct comparisons between immersive VR and low-cost distraction methods during pediatric wound care remain limited.

This study is designed as a single-center, parallel-group randomized controlled trial conducted in the pediatric emergency department of Agri Training and Research Hospital in Turkey. Children aged 5-10 years who require open wound care, including cleansing, dressing, or suturing, are eligible to participate. Following informed consent from parents or guardians and assent from children, participants are randomly allocated in a 1:1:1 ratio to one of three groups: standard wound care alone (control group), standard care with distraction game cards, or standard care with immersive virtual reality glasses.

All participants receive wound care according to institutional clinical protocols. Children in the virtual reality group wear VR glasses displaying age-appropriate immersive content throughout the procedure. Children in the game card group engage with illustrated distraction cards facilitated by a trained researcher. Psychological outcomes, including fear, state anxiety, and pain, are assessed immediately before and shortly after the procedure using validated child-appropriate scales. Physiological responses, including heart rate and peripheral oxygen saturation, are measured concurrently using a pulse oximeter.

The primary objective of the study is to compare post-procedural fear, anxiety, and pain levels between groups. Secondary objectives include evaluation of within-group changes and comparison of physiological stress indicators across interventions. By directly comparing immersive virtual reality with a simple, low-cost distraction method, this study aims to provide clinically relevant evidence to inform the selection of effective, feasible, and scalable non-pharmacological interventions for pediatric wound care.

ELIGIBILITY:
Inclusion Criteria:Children aged 5 to 10 years.

Presentation with an open wound requiring wound care procedures such as cleansing, dressing, debridement, and/or suturing.

Hemodynamic stability at baseline (peripheral oxygen saturation ≥95% and heart rate within age-appropriate limits).

Ability to communicate sufficiently to complete study assessments.

Provision of written informed consent by a parent or legal guardian.

Provision of verbal assent by the child. -

Exclusion Criteria:Presence of neurodevelopmental disorders or communication impairments that could interfere with study assessments.

Significant visual or hearing impairment.

Head or facial wounds that prevent the use of virtual reality glasses.

History of motion sickness or previous adverse reactions to virtual reality.

Receipt of sedatives or systemic opioid analgesics within 6 hours prior to the procedure.

Requirement for procedural sedation during wound care.

Any clinical condition deemed by the attending physician to make participation inappropriate.

-

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Procedural Fear | Immediately before the procedure and within 5 minutes after completion of wound care
  Children's fear related to the wound care procedure, assessed using the Children's Fear Scale. Scores range from 0 (no fear) to 4 (extreme fear), with higher scores indicating greater fear.
Procedural Anxiety | Immediately before the procedure and within 5 minutes after completion of wound care
  Children's state anxiety during wound care, measured using the State Anxiety Inventory for Children. Total scores range from 20 to 60, with higher scores indicating greater anxiety.
Procedural Pain Intensity | Immediately before the procedure and within 5 minutes after completion of wound care
  Pain intensity experienced by children during wound care, assessed using the Wong-Baker Faces Pain Scale. Scores range from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Heart Rate | Immediately before the procedure and within 5 minutes after completion of wound care
  Physiological stress response measured as heart rate (beats per minute) using a fingertip pulse oximeter during a stable 30-second recording period.
Peripheral Oxygen Saturation (SpO₂) | Immediately before the procedure and within 5 minutes after completion of wound care
  Physiological response measured as peripheral oxygen saturation (%) using a fingertip pulse oximeter during a stable 30-second recording period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ağrı Training and Research Hospital, Merkez, AĞRI, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves a pediatric population and was conducted at a single center with a relatively small sample size, which increases the risk of participant re-identification. In addition, the informed consent obtained from parents or guardians did not include permission for data sharing beyond the research team. De-identified aggregate data are reported in the published results.

REFERENCES:
- [Background] Kaya M, Karaman Ozlu Z. The effect of virtual reality on pain, anxiety, and fear during burn dressing in children: A randomized controlled study. Burns. 2023 Jun;49(4):788-796. doi: 10.1016/j.burns.2022.06.001. Epub 2022 Jun 9. PMID 35753857
- [Background] Olbrecht VA, O'Conor KT, Williams SE, Boehmer CO, Marchant GW, Glynn SM, Geisler KJ, Pickerill HM, Ding L, Yang G, King CD. Transient Reductions in Postoperative Pain and Anxiety with the Use of Virtual Reality in Children. Pain Med. 2021 Nov 26;22(11):2426-2435. doi: 10.1093/pm/pnab209. PMID 34175959
- [Background] Thybo KH, Friis SM, Aagaard G, Jensen CS, Dyekjaer CD, Jorgensen CH, Walther-Larsen S. A randomized controlled trial on virtual reality distraction during venous cannulation in young children. Acta Anaesthesiol Scand. 2022 Oct;66(9):1077-1082. doi: 10.1111/aas.14120. Epub 2022 Aug 11. PMID 35898121
- [Background] Sanchez-Caballero E, Ortega-Donaire L, Sanz-Martos S. Immersive Virtual Reality for Pain and Anxiety Management Associated with Medical Procedures in Children and Adolescents: A Systematic Review. Children (Basel). 2024 Aug 13;11(8):975. doi: 10.3390/children11080975. PMID 39201910
- [Background] Addab S, Hamdy R, Thorstad K, Le May S, Tsimicalis A. Use of virtual reality in managing paediatric procedural pain and anxiety: An integrative literature review. J Clin Nurs. 2022 Nov;31(21-22):3032-3059. doi: 10.1111/jocn.16217. Epub 2022 Jan 23. PMID 35068011